CLINICAL TRIAL: NCT06977737
Title: A Phase 1-2 Master Protocol to Study Intravenous ATTR-01 in Adult Participants With Select Epithelial Solid Tumours Under Multiple Sub-protocols
Brief Title: A Study of ATTR-01 in Participants With Select Epithelial Solid Tumours
Acronym: ATTEST
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Accession Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATTR-01-01; ISRCTN38972074 (Registry Identifier: ISRCTN); 1010660 (Other: IRAS)
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental)
  Interventions: Drug: ATTR-01

INTERVENTIONS:
Drug: ATTR-01 — Intravenous injection

SUMMARY:
ATTR-01 is the experimental drug being studied in the ATTEST clinical trial. The drug is made from a common cold virus that has been changed to only infect and multiply in cancer cells. This virus delivers an immune therapy drug into the cancer that is intended to promote a participant's own immune system to attack the cancer. The first part of this trial (sub-protocol A) is a phase 1 trial including dose escalation and expansion at one or more doses. It is the first time that ATTR-01 will be given to humans. If an optimal dose is identified, additional sub-protocols will be added by to further elicit whether ATTR-01 may successfully treat cancer. Expanded access is not available.

ELIGIBILITY:
Inclusion Criteria:

* Consenting male and female adults (18 years of age) with select solid epithelial tumour indications known to have high frequency (75 percent) of αvβ6 integrin receptor expression as detailed in the applicable SP.
* Received and failed/intolerant of Standard of Care (SoC) therapy where eligible (not including neoadjuvant).
* Tumour lesion (not previously irradiated), suitable for safe pre- and post-treatment biopsies.
* Measurable disease by Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Minimum life expectancy anticipated to be greater than three months
* Willing to undertake appropriate measures of hygiene to prevent any spread of virus and protection of vulnerable individuals.
* Adequate organ function.
* Compliant with requirements for prior treatment washout and contraceptive measures applicable to genetically modified organisms (GMOs) and cancer therapies
* Prior immune checkpoint antibody therapies as single agents or in combination with other anti-cancer agents is permissible.

Exclusion Criteria:

* Significant degree of fibrotic disease, including autoimmune diseases (e.g. systemic lupus, rheumatoid arthritis) or idiopathic and occupation-related pulmonary fibrosis.
* Known prior history of intolerance to anti-programmed cell death protein 1 (PD-1) and/or anti-PD-L1 immunotherapy due to toxicity.
* Has any of the comorbid conditions listed in the detailed protocol exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
• Incidence of treatment emergent adverse events (AEs) [safety and tolerability] | 1 year, 2 years and 5 years
• Determination of the optimal dose of ATTR-01 | 1 year, 2 years and 5 years
  • Incidence of AEs, serious adverse events (SAEs), dose limiting toxicities (DLTs), discontinuation of investigational product(s) due to toxicity and clinically significant alterations in vital signs or other clinical safety assessments
• Objective Response Rate (ORR) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
Duration of Response (DoR) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
  From first scan onwards
Time To Response (TTR) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
  From first scan onwards
Progression Free Survival (PFS) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
  From first scan onwards
Overall Survival (OS) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
  From first scan onwards
Maximum reduction in tumour size [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
  From first scan onwards
Duration of Response (DoR) [Evaluation of the anti-tumour activity of ATTR-01 per RECIST V1.1] | 1 year, 2 years and 5 years
  From first scan onwards
To evaluate the viral persistence of ATTR-01 | 1 year
  ATTR-01 viral persistence/blood concentrations
To evaluate the immunogenicity of ATTR-01 | 1 year
  Immunogenicity/Anti-ATTR-01-antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Hardev Pandha, Professor, Study Director — Accession Therapeutics
Locations (7):
- Spain (3):
  - START Barcelona, Barcelona
  - Start Fjd, Madrid
  - Start Hm Ciocc, Madrid
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Cancer Centre, Cardiff, Wales
  - , St James' University Hospital, Leeds
  - Churchill Hospital, Oxford